CLINICAL TRIAL: NCT05918276
Title: Exploratory Clinical Study of Orelabrutinib in Combination With BG Regimen in Patients With Naive and Unfit CLL/SLL Without 17p- or TP53 Mutations
Brief Title: Clinical Study of Orelabrutinib Combined With BG Regimen First-line Treatment of CLL/SLL
Acronym: CLL-OBG
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-202
Record Dates: First submitted 2023-06-08; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: CLL/SLL
Keywords: Orelabrutinib; bendamustine; obintuzumab
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OBG (Experimental)
  Interventions: Drug: Orelabrutinib and BG

INTERVENTIONS:
Drug: Orelabrutinib and BG — Drug: Orelabrutinib Orelabrutinib 200mg, po, qd，C2-C7. Twenty-eight days for a cycle.
  Drug: BG Bendamustin 70mg/m2, IV, d2&d3 inC1, and then d1&d2 inC2-6.Twenty-eight days for a cycle.
  Obintuzumab 100mg IV, d1, 900mg d2, 1000mg d8&d15 in C1, and then 1000mg/m2 IV, d1 in C2-6. Twenty-eight days for a cycle.
  Other Names: OBG

SUMMARY:
This study aims to investigate the treatment of navie CLL/SLL with orelabrutinib, bendamustine and obinutuzumab . The primary endpoint is the rate of CR and uMRD, and the second endpoints are survival time (OS and PFS) and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older or between 18 and 65 years of age with severe illness (non-CLL/SLL associated CIRS ≥ 6);
* ECOG performance status (PS) level 0~2；
* Expected survival is not less than 12 weeks;
* Chronic lymphocytic leukemia/small lymphocytic lymphoma diagnosed by flow cytometry or histopathology according to IWCLL2008 criteria, and CD20 positive;
* Meet at least 1 indication for treatment according to IWCLL2008 criteria or Chinese CLL/SLL guidelines 2022
* Enhanced computed tomography/magnetic resonance imaging (CT/MRI) to detect measurable lesions: at least one lymph node with a maximum axis of more than 1.5 cm and one measurable vertical dimension; for patients with chronic lymphocytic leukemia, only peripheral circulating lymphocyte count must be > 5000/μL (or 5×10^9/L);
* Have not received systematic treatment for CLL/SLL in the past;
* The main organs are functioning normally, the following criteria are met:

  1. Routine blood test standards should meet:

     Absolute neutrophil (ANC) ≥1.0×109/L, platelet (PLT) ≥30×109/L; unless bone marrow and hematopoietic insufficiency is confirmed to be due to CLL/SLL
  2. Biochemical examination should meet the following standards:

     1. TBIL<2.0× ULN, CLL/SLL liver involvement or confirmed Gilbert syndrome (normal direct bilirubin), total bilirubia ≤ 3 times ULN;
     2. ALT and AST <2.5×ULN (ALT and AST <5×ULN for CLL/SLL liver involvement);
     3. Endogenous creatinine clearance ≥ 30 ml/min (Cockcroft-Gault formula).
* Women of childbearing age must have taken reliable contraceptive measures or have taken a pregnancy test (serum or urine) within 7 days prior to enrollment, have a negative result, and be willing to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the test drug. For men, consent to appropriate methods of contraception or surgical sterilization during the trial and 8 weeks after the last administration of the test drug must be agreed;
* Subjects voluntarily join the study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Patients with 17P- chromosome abnormalities or TP53 mutations;
* Current or previous biopsy pathology confirms conversion to Richter's syndrome;
* Have active and uncontrolled autoimmune cytopenias, including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura;
* Patients with central nervous system invasion;
* Glucocorticoid therapy (at a dose equal to or greater than 20 mg/day of prednisone or equivalent) within 14 days prior to the first dose, excluding inhalation, topical medication, intra-articular medication, and prophylaxis before or after iodine contrast use; After discussion with the team leader, higher doses, longer steroid therapy may be allowed in the following cases:

  1. treatment of autoimmune hemolysis or autoimmune thrombocytopenia associated with CLL/SLL disease;
  2. Acute exacerbations due to short-term (within 14 days) use of inactive infections for diseases not associated with CLL/SLL (e.g., arthritis, asthma), including steroid dose adjustment required for adrenal insufficiency;
* Previous or concurrent uncured malignant tumors, except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and superficial bladder cancer;
* Suffering from the following cardiovascular diseases: grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval QTc >480ms); According to NYHA standards, grade III.~IV. cardiac insufficiency, or cardiac ultrasound showed left ventricular ejection fraction (LVEF) < 50%;
* Coagulation dysfunction (INR>1.5 or prothrombin time (PT) >ULN+4 seconds or APTT >1.5 ULN), bleeding tendency or receiving thrombolysis or anticoagulation therapy;
* Arteriovenous thrombotic events that occurred within 12 months before enrollment, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
* Known hereditary or acquired bleeding and thrombosis (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.);
* Have undergone major surgical procedures or developed severe traumatic injuries, fractures or ulcers within 4 weeks of enrollment;
* Factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction;
* Active infection requiring antimicrobial therapy (such as antibacterial drugs and antiviral drugs, excluding chronic hepatitis B anti-hepatitis B treatment and antifungal treatment);
* Active hepatitis B (HBV DNA≥2000 IU/mL or 10000 copy number/mL) or hepatitis C (positive for hepatitis C antibodies and HCV RNA above the lower limit of the assay);
* Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
* Have participated in clinical trials of other antitumor drugs within 4 weeks before enrollment;
* Those who have received strong CYP3A4 inhibitor therapy within 7 days before enrollment, or received strong CYP3A4 inducer therapy within 12 days before participating in the study;
* Pregnant or lactating women; Patients of childbearing potential who are unwilling or unable to use effective contraception; 19. Other circumstances that may affect the conduct of clinical research and the determination of research results as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of CR and uMRD | Approximately 2 years.
  The proportion of patients with CR and undetectable peripheral blood/bone marrow minimal residual disease in the end of combination therapy. Patients with CRi are counted as CR.

SECONDARY OUTCOMES:
The rate of CR/CRu and uMRD | Approximately 2 years.
  The proportion of patients with CR/CRu and undetectable peripheral blood/bone marrow minimal residual disease in the end of combination therapy. Patients with CRi are counted as CR. CRu is defined as a large spleen size of 16cm or less, and the rest of the indicators meet CR/CRi standards.
The Rate of uMRD | Approximately 2 years.
  According to the detection of Shihe Gene [igNGS kit], no residual leukemia cells were detected in a million peripheral blood or bone marrow cells.
PFS（progression-free survival） | Up to 8 years.
  Progression-free survival (PFS) is defined as the time from the date of first administration to the date of first disease progression or death from any cause, whichever occurs first.
OS（overall survival） | Up to 10 years.
  Overall survival (OS) refers to the time from receiving the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ru Feng, Master, Study Chair — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - The Central Hospital Of Wuan, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan